CLINICAL TRIAL: NCT02688374
Title: A Single-Dose, Open-Label, Three-way Crossover Bioequivalence Study of Three, 2 mg Nicotine Chewing Gums (Two Tests and One Reference) in Chinese Male Healthy Adult Smokers
Brief Title: A Bioequivalence Study of Three, 2 mg Nicotine Chewing Gums (Two Tests and One Reference) in Healthy Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 204979
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

ARMS (6):
- Treatment A:Treatment B:Treatment C (Other): Participants will be administered with Treatment A(Nicorette 2 mg coated mint gum) followed by Treatment B (Nicotinell 2 mg coated mint gum) followed by Treatment C (Nicotinell 2 mg coated fruit flavor gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum
- Treatment B:Treatment C:Treatment A (Other): Participants will be administered with Treatment B (Nicotinell 2 mg coated mint gum) followed by Treatment C (Nicotinell 2 mg coated fruit flavor gum) followed by Treatment A(Nicorette 2 mg coated mint gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum
- Treatment C:Treatment A:Treatment B (Other): Participants will be administered with Treatment C (Nicotinell 2 mg coated fruit flavor gum) followed by Treatment A(Nicorette 2 mg coated mint gum) followed by Treatment B (Nicotinell 2 mg coated mint gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum
- Treatment A: Treatment C:Treatment B (Other): Participants will be administered with Treatment A (Nicorette 2 mg coated mint gum) followed by Treatment C (Nicotinell 2 mg coated fruit flavor gum) followed by Treatment B (Nicotinell 2 mg coated mint gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum
- Treatment B:Treatment A: Treatment C (Other): Participants will be administered with Treatment B (Nicotinell 2 mg coated mint gum) followed by Treatment A (Nicorette 2 mg coated mint gum) followed by Treatment C (Nicotinell 2 mg coated fruit flavor gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum
- Treatment C:Treatment B:Treatment A (Other): Participants will be administered with Treatment C (Nicotinell 2 mg coated fruit flavor gum) followed by Treatment B (Nicotinell 2 mg coated mint gum) followed by Treatment A (Nicorette 2 mg coated mint gum). Administration of each treatment will be separated by clinical furlough period of at least 7 days and not more than 10 days.
  Interventions: Other: Treatment A: Nicorette 2 mg coated mint gum; Other: Treatment B: Nicotinell 2 mg coated mint gum; Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum

INTERVENTIONS:
Other: Treatment A: Nicorette 2 mg coated mint gum — Participants will be administered with 2 mg coated mint gum of Nicorette
Other: Treatment B: Nicotinell 2 mg coated mint gum — Participants will be administered with 2 mg coated mint gum of Nicotinell
Other: Treatment C: Nicotinell 2 mg coated fruit flavor gum — Participants will be administered with 2 mg coated fruit flavor gum of Nicotinell

SUMMARY:
This is a randomized, open-label, single-dose, three-period, crossover, single-center comparative bioavailability (BA) study under fasting condition in Chinese healthy male adult participants with a history of cigarette smoking. The participants will be admitted to the investigational clinic at least 38 hours before dosing and will remain domiciled until the completion of all study procedures at approximately 24 hours after dosing. Three toothpastes (one is commercial non-medicated non-nicotine containing chewing gum and other two are nicotine containing gums) will be provided across the 3 treatment periods. During each of the 3 treatment periods, participants will be under supervision in a non-smoking area and will abstain from smoking.There will be a total of at least 7 days and not more than 10 days (clinical furlough period) between treatment periods. Twenty (20) blood samples will be collected for pharmacokinetic (PK) analysis at baseline and multiple time points following study drug administration. The trial duration will be approximately 49 days and up to 55 days from screening to study end including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand and provide written informed consent before any assessment is performed, understand the study procedures, and be willing to complete the required assessments and the study.
* Chinese male participants between 18 and 45 years of age (inclusive) in general good physical health as judged by the Investigator.
* Normal vital signs as follows:
* Oral body temperature between 35.0 and 37.5 ºC (95 and 99.5 F) inclusive
* Supine systolic blood pressure between 90 and 140 mmHg inclusive
* Supine diastolic blood pressure between 55 and 90 mmHg inclusive
* Pulse rate between 50 and 100 beats per minute (bpm) inclusive
* History of cigarette smoking of at least 10 cigarettes per day continuously for the past 3 months prior to screening.
* Body weight ≥ 50 kg, Body Mass Index (BMI) between 19 and 28 at screening.
* Ability to communicate and comply with all study requirements including the study specific chewing and swallowing procedures.

Exclusion Criteria:-

* Use of other investigational drugs within 30 days or 10 half-lives of enrollment, whichever is longer.
* History of or known hypersensitivity to the study drug or excipients.
* Diagnosis of long QT syndrome or QTc > 450 msec for males at screening.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance.
* History of malignancy or neoplastic disease of any organ system treated or untreated, orthostatic hypotension, cardiovascular disease, stroke, TIA, fainting or blackouts, clinically significant metabolic, pulmonary, neurological, hematological, autoimmune, psychiatric or endocrine disorders.. within the past 5 years prior to screening.
* Any evidence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinological, metabolic, autoimmune, neurological, psychiatric, other diseases or other clinically significant laboratory findings at screening.
* Participant has used any medication within two weeks before first scheduled study drug administration or within less than 10 times the elimination half-life of the respective drug.
* Unable to comply with the chewing and/or swallowing rhythm requirements (> 5% deviation of the total counts over 30 minutes) after trying either one of the two training sessions for 3 times.
* CO > 12 ppm after at least 38 hours confinement period in clinics prior to first dosing.
* Participants reports consumption of any drug metabolizing enzyme inducing or inhibiting aliments, evidence of current alcohol abuse or reports consumption exceeding 35 g of pure alcohol per day.
* Any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis, positive results in any of the virology tests for Human immunodeficiency virus (HIV)-Ab, Hepatitis C virus (HCV)-Ab, Surface antigen of the hepatitis B virus (HBs-Ag), and Tp-Ab.
* Participation in a previous clinical study with or without another investigational product and with ~470 ml blood drawn, or blood donation within the last 3 months prior to screening or previous enrollment into the current study.
* Vulnerable individual
* Inability to be venipuncture and/or tolerate venous access, unwilling to accept slight irritation of the throat and increased salivation due to nicotine gum administration.
* Unable or unwilling to discontinue the use or consumption of cigarette smoking, any nicotine containing products, Oral, local or topical pharmaceutical agents, consumption of caffeine/theophylline - containing products, grapefruit, Seville orange, orange, lemon, lime, apple, and pineapple, performance of unaccustomed strenuous physical exercise.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-06-12 (Actual); Study Completion 2016-06-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to last sampling time [AUC(0-t)] | 2 days
  AUC(0-t) will be calculated using the trapezoidal rule. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Area under the curve from time zero extrapolated to infinity [AUC(0-inf)] | 2 days
  The area under the plasma concentration versus time curve will be calculated from time 0 to infinity where AUC = AUClast + Clast/λz Clast is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Maximum plasma concentration (Cmax) | 2 days
  Cmax will be obtained graphically from the plasma concentration over time profile. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Time to reach maximum plasma concentration (Tmax) | 2 days
  Tmax will be obtained graphically from the plasma concentration over time profile. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Termination rate constant (Lambda_z) | 2 days
  Lambda_z will be computed as the slope of the regression line of ln (C(t)) on time. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Elimination half life (t1/2) | 2 days
  T1/2 will be computed as T1/2 = 0.693/ λz. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Systemic clearance (CL/F) | 2 days
  CL/F will be calculated as the Dose/AUCinf, where Dose is the actual nicotine dose released. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.
Apparent volume of distribution (Vd/F) | 2 days
  Vd/F will be determined by the following equation: Vz/F = Dose/(lambda_z · AUCinf), where Dose is the actual nicotine dose released. Twenty (20) blood samples will be collected at baseline and multiple timepoints following study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China